CLINICAL TRIAL: NCT06982391
Title: CompACT: A Program for Enhancing Compassion, Social Support, Psychological Flexibility, and Resilience in Female Breast Cancer Survivors
Brief Title: Compassion, Social Support, Flexibility, and Resilience Program for Women Surviving Breast Cancer
Acronym: ReACT
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Ela Ari, Assistant Professor, Medipol University
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 1357-2481
Record Dates: First submitted 2025-05-13; First posted 2025-05-21 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Breast Cancer Survivor; Mastectomy
Keywords: resilience; psychological flexibility; values; self as compassionate context; social support; value-driven committed action; acceptance; defusion

STUDY DESIGN:
Intervention Model Description: An interventional study design for a single group typically involves selecting a group of participants who meet specific inclusion criteria, and then applying an intervention to this group. The participants are assessed before the intervention (pre-test), followed by the application of the intervention, which could be a treatment, educational program, or behavioral change activity. After the intervention, participants are assessed again (post-test) to evaluate any changes in the targeted outcomes. The design includes a follow-up period to assess the sustainability of the effects. The focus of a two arms randomized control design is on examining the impact of the intervention on the group, with comparisons made between pre- and post-intervention measurements and the standard care group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- This is the intervention arm (Experimental): Participants assigned to the intervention arm will take part in the Resilience-Focused Acceptance and Commitment Therapy (ReACT) program. This program includes three weekly 90-minute structured group sessions specifically designed for women who have undergone mastectomy following breast cancer. The intervention integrates core Acceptance and Commitment Therapy (ACT) techniques (acceptance, cognitive defusion, mindfulness, values clarification, committed action) with a focus on psychological resilience and enhancing perceived social support. Participants will also engage in experiential exercises and home practices aimed at improving psychological flexibility, coping skills, and post-cancer adjustment.
  Interventions: Behavioral: Resilience-Focused Acceptance and Commitment Therapy (ReACT) Program
- Control Arm (Experimental): This group will receive standard care
  Interventions: Other: No intervention

INTERVENTIONS:
Behavioral: Resilience-Focused Acceptance and Commitment Therapy (ReACT) Program — The Resilience-Focused Acceptance and Commitment Therapy (ReACT) program is a structured, group-based psychological intervention specifically designed for women who have undergone mastectomy following breast cancer. The program consists of three weekly 90-minute sessions integrating core ACT processes, including acceptance, defusion, mindfulness, values clarification, and committed action, with an emphasis on building psychological resilience, self-compassion, and enhancing perceived social support. The program uniquely combines evidence-based ACT techniques with group exercises focused on post-cancer psychosocial adjustment.
  Arms: This is the intervention arm
Other: No intervention — Standard Care
  Arms: Control Arm

SUMMARY:
The goal of this clinical trial is to investigate the effects of an Acceptance and Commitment Therapy (ACT) based program (ReACT) to increase social support, compassion and psychological flexibility on psychological resilience in women undergoing mastectomy. The main question it aims to answer is: Does the ReACT program improve participants' resilience by increasing social support, compassion, and psychological flexibility? Researchers will compare intervention group to control group to see if ReACT program works to improve participants' resilience.

Researchers will randomly divide participants into two groups: intervention group and control group.

* Participants will complete some questionnaires.
* Participants in the intervention group will join a 3-week ACT-based psychological flexibility program. This program consists of sessions that last 90 minutes each. The program adopts the core principles of ACT and aims to help participants develop skills in mindfulness, acceptance, value-driven living, and cognitive defusion.
* Participants will complete the same questionnaires again after the program.
* Participants will complete the same questionnaires again 1 month after the program ends.

DETAILED DESCRIPTION:
Intervention studies aiming to increase psychological resilience in women with breast cancer after mastectomy are gaining increasing attention in the literature. Various studies highlight the positive effects of social support and psychological flexibility on the mental health of cancer patients. In particular, social support enhances the stress-coping capacity of cancer patients and strengthens their psychological resilience (Hulbert-Williams et al., 2015).

Acceptance and Commitment Therapy (ACT)-based interventions are considered an effective approach for coping with chronic illnesses. Studies on cancer patients emphasize that ACT increases psychological flexibility, helping patients accept challenging emotions and focus on meaningful areas of life (Hayes et al., 2006).

The innovative aspect of this study is the evaluation of both social support and ACT-based flexibility interventions together, examining their combined effects on psychological resilience after breast cancer. Research that comprehensively explores the interaction between social support and psychological flexibility remains limited. This study offers a more effective model for enhancing resilience in cancer patients by assessing the combined impact of components such as social support and psychological flexibility.

In this context, the research contributes significantly to the literature by presenting an integrated approach to increasing psychosocial resilience in the post-breast cancer period and offering a new perspective for intervention studies in this field.

The study includes a total of 20 female participants, aged between 18 and 65, who have undergone mastectomy and voluntarily agree to participate. Participation is voluntary, and participants may withdraw at any time without consequence.

The following scales are used in the study: Sociodemographic and Clinical Information Form, Interpersonal Support Evaluation List-12 (ISEL-12), Self-Compassion Scale-Short Form (SCS-SF), Acceptance and Action Questionnaire-II (AAQ-II), Brief Resilience Scale (BRS), and PROMIS Scales - Global Health Scale, Social Roles and Activities Participation - Short Form 4a, Depression - Short Form 4a, Anxiety - Short Form 4a.

Program Sessions

Session 1: Introduction, Introduction to ReACT Program Purposes, ReACT Matrix, Identifying Values, Defusion

Goal: Introduce the program to participants. They explore their values using the Matrix, identify thoughts that distance them from their values, explore their behaviors, focus to observe their thoughts, practice a present moment awareness exercise, and learn cognitive defusion.

Content:

Psychoeducation: Discuss the importance of psychological resilience, social support, and compassion after breast cancer (Hayes et al., 2006).

Exercise: Participants practice the "Present Moment Exercise" to ground themselves in the here and now with openness and awareness. This practice helps them observe thoughts without becoming entangled in them, supporting more intentional and values-based actions.

Session 2: Acceptance of Anxiety, Compassion, and Action

Goal: Help participants manage difficult emotions and understand how they can move forward while accepting difficult emotions.

Content:

Psychoeducation: Participants explore the questions "What are emotions?" and "What is the function of emotions?" They learn that emotions serve as signals of what matters in life. The idea of making space for emotions instead of fighting them is introduced, along with the insight that this can help reveal underlying values. The link between emotions and values is explored with examples.

Exercise: The sky metaphor is introduced to support acceptance of difficult emotions. If it is not effective, an alternative acceptance exercise is offered.

Session 3: Value-Driven Actions, Sustainability, and Committed Action Toward Receiving and Giving Compassion

Goal: Explore values, value-oriented behaviors, and action planning related to giving and receiving compassion.

Content:

Action Plan: Participants identify daily behaviors that align with their values and develop an action plan (Moreno et al., 2022).

Group Sharing: Participants share their experiences and what they have learned throughout the sessions (Hayes et al., 2006).

Exercise: Participants receive a guide to monitor their progress and maintain value-driven actions (Kabat-Zinn, 1990).

Monitoring and Evaluation

Goal: Evaluate the effects of the intervention and support sustainability.

Content:

Post-Program Evaluation: Final assessments are conducted immediately after the program ends.

Follow-Up: A Zoom group monitoring session is held four weeks later.

Review: During follow-up, changes in psychological resilience, psychological flexibility, compassion, value-based living, and PROMIS scales are reviewed (Neff, 2003; Moreno et al., 2022).

ELIGIBILITY:
Inclusion Criteria:

* Female participants aged between 18 and 65 years.
* Participants who have undergone a mastectomy.
* Participants who voluntarily agree to participate in the study.

Exclusion Criteria:

-

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female individuals who have had a mastectomy
Enrollment: 20 (Estimated)
Dates: Start 2025-04-12 (Actual); Primary Completion 2026-01-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
Resilience | three weeks
  Psychological resilience will be assessed using the Brief Resilience Scale (BRS). The outcome will measure changes from baseline (pre-intervention) to post-intervention (immediately after the 3-week program). The Brief Resilience Scale evaluates the individual's ability to recover from stress and adversity.

SECONDARY OUTCOMES:
Self Compassion | three weeks
  Self-compassion will be assessed using the Self-Compassion Scale - Short Form (SCS-SF). The outcome will measure changes from baseline (pre-intervention) to post-intervention (immediately after the 3-week program). The SCS-SF evaluates an individual's ability to treat themselves with kindness, understanding, and non-judgmental awareness during times of difficulty or failure.
Psychological Flexibility | Three weeks
  Psychological flexibility will be assessed using the Acceptance and Action Questionnaire-II (AAQ-II). The outcome will measure changes from baseline (pre-intervention) to post-intervention (immediately after the 3-week program). The AAQ-II evaluates an individual's ability to accept difficult thoughts and feelings without unnecessary struggle and to engage in values-based actions despite internal discomfort.
Well-being | Three weeks
  Overall well-being and quality of life will be assessed using the PROMIS Global Health Scale. The outcome will measure changes from baseline (pre-intervention) to post-intervention (immediately after the 3-week program). The PROMIS Global Health Scale evaluates physical, mental, and social health to provide a comprehensive picture of an individual's perceived general health and life satisfaction.

CONTACTS AND LOCATIONS:
Overall Officials: Ela Arı, Assistant Professor, Principal Investigator — Medipol University
Locations (1):
- Florence Nightingale Hospital, Istanbul, Turkey (Türkiye)